CLINICAL TRIAL: NCT03014167
Title: Field Studies on the Feasibility of Interrupting the Transmission of Soil-transmitted Helminths (STH) DeWorm3 Project
Brief Title: Field Studies on the Feasibility of Interrupting the Transmission of Soil-transmitted Helminths (STH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Imperial College London (Other); London School of Hygiene and Tropical Medicine (Other); Institut de Recherche Clinique du Bénin (IRCB) (Unknown); Institut de Recherche pour le Developpement (Other Government); Christian Medical College, Vellore, India (Other); Blantyre Institute for Community Ophthalmology (BICO) (Unknown); Swiss Tropical & Public Health Institute (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Judd Walson, Professor in Departments of Global Health, Medicine (Infectious Disease), Pediatrics and Epidemiology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000180; 1R01AI155739-01A1 (NIH)
Record Dates: First submitted 2016-12-30; First posted 2017-01-09 (Estimated); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-07

CONDITIONS: Helminthiasis; Filariasis
Keywords: transmission interruption; intestinal nematodes; soil-transmitted helminths; mass drug administration; Benin; India; Malawi
MeSH Terms: conditions — Helminthiasis; Filariasis | interventions — Albendazole

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Mass drug administration intervention is not blinded to study participants but investigators and outcome assessors remain blind to link between allocation and outcome data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Community-wide deworming (Experimental): Twice-yearly community-wide treatment delivered by drug distributors door to door or via community gatherings, depending upon the format of the prior LF program, for three years. All individuals above the age of 12 months will receive a single dose of albendazole.
  Interventions: Drug: Albendazole
- Targeted deworming (Active Comparator): Pre-school (pre-SAC) and school-age children (SAC) 12 months of age and older will receive albendazole delivered in accordance with national Ministry of Health guidelines for three years.
  Interventions: Drug: Albendazole

INTERVENTIONS:
Drug: Albendazole — All eligible individuals will receive a single dose of 400 mg albendazole.
  Other Names: Albenza

SUMMARY:
Over 1.5 billion people are infected with soil-transmitted helminths (STH). Global STH guidelines recommend MDA (mass drug administration) of albendazole or mebendazole to targeted populations, including pre-school age children and school-age children. However mathematical models suggests that current MDA strategies are not sufficient for interrupting disease transmission in most areas. Meanwhile many lymphatic filariasis (LF) programs have successfully treated entire populations with albendazole (in combination with ivermectin or diethylcarbamazine) and are transitioning to a state of post-MDA surveillance. This project will conduct a series of community-based cluster randomized trials in India, Malawi, and Benin to determine if maintaining three years of MDA with albendazole to entire communities following the cessation of LF programs can interrupt STH transmission in focal geographic areas. Additionally, this study aims to compare the efficacy of community-wide MDA versus targeted MDA of children in interrupting the transmission of STH. Nested implementation science research will be used to optimize the intervention, identify contextual factors influencing trial efficacy, and evaluate the feasibility of sustaining and scaling community-wide MDA for STH. These data will provide evidence necessary to inform future guidelines, policies, and operational plans as country partners engage in intensified approaches to eliminate these disabling diseases.

ELIGIBILITY:
Treatment Inclusion Criteria:

* Ages 12 months and older

Treatment Exclusion Criteria:

* Children under 12 months of age
* Pregnant women in their first trimester
* History of adverse reaction to benzimidazoles

Outcome Sampling Inclusion Criteria:

* Resident of study clusters
* Ages 12 months and older
* Willingness of adult aged 18 years and above (or age as per country specific ethical guidelines) or parent/guardian of child to provide written informed consent
* Provision of written assent to participate from children aged 8 years and above (or age as per country specific ethical guidelines)

Outcome Sampling Exclusion Criteria:

* Less than 12 months of age
* Individuals who do not typically reside in the study cluster
* Nonconsenting or assenting individuals, as applicable

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 357716 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judd L Walson, MD, MPH, Principal Investigator — University of Washington, Departments of Global Health, Medicine (Infectious Disease), Pediatrics and Epidemiology
Locations (3):
- Institut de Recherche pour le Développement, Comé, Benin
- Christian Medical College, Vellore, India
- London School of Hygiene and Tropical Medicine, Mangochi, Malawi

REFERENCES:
- [Derived] Ajjampur SSR, Aruldas K, Asbjornsdottir KH, Avokpaho E, Bailey R, Cottrell G, Galagan SR, Halliday KE, Houngbegnon P, Ibikounle M, Israel GJ, Kaliappan SP, Kalua K, Legge H, Littlewood DTJ, Luty AJF, Manuel M, Massougbodji A, Means AR, Oswald WE, Pilotte N, Pullan R, Ramesh RM, Samikwa L, Simwanza J, Thomas KK, Williams SA, Witek-McManus S, Walson JL; DeWorm3 Trials Team. Feasibility of interrupting the transmission of soil-transmitted helminths: the DeWorm3 community cluster-randomised controlled trial in Benin, India, and Malawi. Lancet. 2025 Aug 2;406(10502):475-488. doi: 10.1016/S0140-6736(25)00766-4. PMID 40752908
- [Derived] Means AR, Asbjornsdottir KH, Sharrock KC, Galagan SR, Aruldas K, Avokpaho E, Chabi F, Halliday KE, Houngbegnon P, Israel GJ, Kaliappan SP, Kennedy D, Legge H, Oswald WE, Palanisamy G, Rogers E, Timothy J, Pearman E, Ramesh RM, Simwanza J, Sheik-Abdullah JF, Sheikh M, Togbevi CI, Witek-McManus S, Pullan RL, Bailey R, Kalua K, Ibikounle M, Luty AJF, Ajjampur SSR, Walson JL. Coverage of community-wide mass drug administration platforms for soil-transmitted helminths in Benin, India, and Malawi: findings from the DeWorm3 project. Infect Dis Poverty. 2024 Oct 8;13(1):72. doi: 10.1186/s40249-024-01241-0. PMID 39380086
- [Derived] Witek-McManus S, Simwanza J, Msiska R, Mangawah H, Oswald W, Timothy J, Galagan S, Pearman E, Shaikh M, Legge H, Walson J, Juziwelo L, Davey C, Pullan R, Bailey RL, Kalua K, Kuper H. Disability in childhood and the equity of health services: a cross-sectional comparison of mass drug administration strategies for soil-transmitted helminths in southern Malawi. BMJ Open. 2024 Sep 5;14(9):e083321. doi: 10.1136/bmjopen-2023-083321. PMID 39242171
- [Derived] Saxena M, Roll A, Walson JL, Pearman E, Legge H, Nindi P, Chirambo CM, Titus A, Johnson J, Belou EA, Togbevi CI, Chabi F, Avokpaho E, Kalua K, Ajjampur SSR, Ibikounle M, Aruldas K, Means AR. "Our desire is to make this village intestinal worm free": Identifying determinants of high coverage of community-wide mass drug administration for soil transmitted helminths in Benin, India, and Malawi. PLoS Negl Trop Dis. 2024 Feb 6;18(2):e0011819. doi: 10.1371/journal.pntd.0011819. eCollection 2024 Feb. PMID 38319937
- [Derived] Kazura E, Johnson J, Morozoff C, Aruldas K, Avokpaho E, Togbevi CI, Chabi F, Gwayi-Chore MC, Nindi P, Titus A, Houngbegnon P, Kaliappan SP, Jacob Y, Simwanza J, Kalua K, Walson JL, Ibikounle M, Ajjampur SSR, Means AR. Identifying opportunities to optimize mass drug administration for soil-transmitted helminths: A visualization and descriptive analysis using process mapping. PLoS Negl Trop Dis. 2024 Jan 4;18(1):e0011772. doi: 10.1371/journal.pntd.0011772. eCollection 2024 Jan. PMID 38175837
- [Derived] Ramesh RM, Oswald WE, Israel GJ, Aruldas K, Galagan S, Legge H, Puthupalayam Kaliappan S, Walson J, Halliday KE, Ajjampur SSR. Representativeness of a mobile phone-based coverage evaluation survey following mass drug administration for soil-transmitted helminths: a comparison of participation between two cross-sectional surveys. BMJ Open. 2023 Oct 29;13(10):e070077. doi: 10.1136/bmjopen-2022-070077. PMID 37899143
- [Derived] Sheahan W, Anderson R, Aruldas K, Avokpaho E, Galagan S, Goodman J, Houngbegnon P, Israel GJ, Janagaraj V, Kaliappan SP, Means AR, Morozoff C, Pearman E, Ramesh RM, Roll A, Schaefer A, Simwanza J, Witek-McManus S, Ajjampur SSR, Bailey R, Ibikounle M, Kalua K, Luty AJF, Pullan R, Walson JL, Asbjornsdottir KH. Overestimation of school-based deworming coverage resulting from school-based reporting. PLoS Negl Trop Dis. 2023 Apr 10;17(4):e0010401. doi: 10.1371/journal.pntd.0010401. eCollection 2023 Apr. PMID 37036890
- [Derived] Aruldas K, Israel GJ, Johnson J, Titus A, Saxena M, Kaliappan SP, Ramesh RM, Walson JL, Means AR, Ajjampur SSR. Impact of adverse events during community-wide mass drug administration for soil-transmitted helminths on subsequent participation-a Theory of Planned Behaviour analysis. PLoS Negl Trop Dis. 2023 Mar 14;17(3):e0011148. doi: 10.1371/journal.pntd.0011148. eCollection 2023 Mar. PMID 36917597
- [Derived] Aruldas K, Dawson K, Saxena M, Titus A, Johnson J, Gwayi-Chore MC, Muliyil J, Kang G, Walson JL, Khera A, Ajjampur SSR, Means AR. Evaluation of opportunities to implement community-wide mass drug administration for interrupting transmission of soil-transmitted helminths infections in India. PLoS Negl Trop Dis. 2023 Mar 10;17(3):e0011176. doi: 10.1371/journal.pntd.0011176. eCollection 2023 Mar. PMID 36897877
- [Derived] Roll A, Saxena M, Orlan E, Titus A, Juvekar SK, Gwayi-Chore MC, Avokpaho E, Chabi F, Togbevi CI, Belou Elijan A, Nindi P, Walson JL, Ajjampur SSR, Ibikounle M, Kalua K, Aruldas K, Means AR. Policy stakeholder perspectives on barriers and facilitators to launching a community-wide mass drug administration program for soil-transmitted helminths. Glob Health Res Policy. 2022 Dec 2;7(1):47. doi: 10.1186/s41256-022-00281-z. PMID 36461087
- [Derived] Morozoff C, Avokpaho E, Puthupalayam Kaliappan S, Simwanza J, Gideon SP, Lungu W, Houngbegnon P, Galactionova K, Sahu M, Kalua K, Luty AJF, Ibikounle M, Bailey R, Pullan R, Ajjampur SSR, Walson J, Means AR. Costs of community-wide mass drug administration and school-based deworming for soil-transmitted helminths: evidence from a randomised controlled trial in Benin, India and Malawi. BMJ Open. 2022 Jul 8;12(7):e059565. doi: 10.1136/bmjopen-2021-059565. PMID 35803632
- [Derived] Avokpaho E, Lawrence S, Roll A, Titus A, Jacob Y, Puthupalayam Kaliappan S, Gwayi-Chore MC, Chabi F, Togbevi CI, Elijan AB, Nindi P, Walson JL, Ajjampur SSR, Ibikounle M, Kalua K, Aruldas K, Means AR. It depends on how you tell: a qualitative diagnostic analysis of the implementation climate for community-wide mass drug administration for soil-transmitted helminth. BMJ Open. 2022 Jun 14;12(6):e061682. doi: 10.1136/bmjopen-2022-061682. PMID 35701056
- [Derived] Avokpaho EFGA, Houngbegnon P, Accrombessi M, Atindegla E, Yard E, Rubin Means A, Kennedy DS, Littlewood DTJ, Garcia A, Massougbodji A, Galagan SR, Walson JL, Cottrell G, Ibikounle M, Asbjornsdottir KH, Luty AJF. Factors associated with soil-transmitted helminths infection in Benin: Findings from the DeWorm3 study. PLoS Negl Trop Dis. 2021 Aug 17;15(8):e0009646. doi: 10.1371/journal.pntd.0009646. eCollection 2021 Aug. PMID 34403424
- [Derived] Means AR, Orlan E, Gwayi-Chore MC, Titus A, Kaliappan SP, Togbevi CI, Chabi F, Halliday KE, Nindi P, Avokpaho E, Kalua K, Ibikounle M, Ajjampur SSR, Weiner BJ, Walson JL, Aruldas K. Structural readiness to implement community-wide mass drug administration programs for soil-transmitted helminth elimination: results from a three-country hybrid study. Implement Sci Commun. 2021 Jul 19;2(1):80. doi: 10.1186/s43058-021-00164-3. PMID 34281614
- [Derived] Galactionova K, Sahu M, Gideon SP, Puthupalayam Kaliappan S, Morozoff C, Ajjampur SSR, Walson J, Rubin Means A, Tediosi F. Costing interventions in the field: preliminary cost estimates and lessons learned from an evaluation of community-wide mass drug administration for elimination of soil-transmitted helminths in the DeWorm3 trial. BMJ Open. 2021 Jul 5;11(7):e049734. doi: 10.1136/bmjopen-2021-049734. PMID 34226233
- [Derived] Witek-McManus S, Simwanza J, Chisambi AB, Kepha S, Kamwendo Z, Mbwinja A, Samikwa L, Oswald WE, Kennedy DS, Timothy JWS, Legge H, Galagan SR, Emmanuel-Fabula M, Schaer F, Asbjornsdottir K, Halliday KE, Walson JL, Juziwelo L, Bailey RL, Kalua K, Pullan RL. Epidemiology of soil-transmitted helminths following sustained implementation of routine preventive chemotherapy: Demographics and baseline results of a cluster randomised trial in southern Malawi. PLoS Negl Trop Dis. 2021 May 12;15(5):e0009292. doi: 10.1371/journal.pntd.0009292. eCollection 2021 May. PMID 33979325
- [Derived] Ajjampur SSR, Kaliappan SP, Halliday KE, Palanisamy G, Farzana J, Manuel M, Abraham D, Laxmanan S, Aruldas K, Rose A, Kennedy DS, Oswald WE, Pullan RL, Galagan SR, Asbjornsdottir K, Anderson RM, Muliyil J, Sarkar R, Kang G, Walson JL. Epidemiology of soil transmitted helminths and risk analysis of hookworm infections in the community: Results from the DeWorm3 Trial in southern India. PLoS Negl Trop Dis. 2021 Apr 30;15(4):e0009338. doi: 10.1371/journal.pntd.0009338. eCollection 2021 Apr. PMID 33930024
- [Derived] DeWorm3 Trials Team. Baseline patterns of infection in regions of Benin, Malawi and India seeking to interrupt transmission of soil transmitted helminths (STH) in the DeWorm3 trial. PLoS Negl Trop Dis. 2020 Nov 2;14(11):e0008771. doi: 10.1371/journal.pntd.0008771. eCollection 2020 Nov. PMID 33137100
- [Derived] Asbjornsdottir KH, Ajjampur SSR, Anderson RM, Bailey R, Gardiner I, Halliday KE, Ibikounle M, Kalua K, Kang G, Littlewood DTJ, Luty AJF, Means AR, Oswald W, Pullan RL, Sarkar R, Schar F, Szpiro A, Truscott JE, Werkman M, Yard E, Walson JL; DeWorm3 Trials Team. Assessing the feasibility of interrupting the transmission of soil-transmitted helminths through mass drug administration: The DeWorm3 cluster randomized trial protocol. PLoS Negl Trop Dis. 2018 Jan 18;12(1):e0006166. doi: 10.1371/journal.pntd.0006166. eCollection 2018 Jan. PMID 29346377
- See also: University of Washington DeWorm3 Website — http://deworm3.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were approached during a baseline census and offered the opportunity to participant in the study. Consent was taken from an adult household member for the entire household.
Pre-assignment Details: Prior to restricted randomization, clusters were demarcated (40 per site) with 1650+ individuals following local administrative boundaries. Study clusters were then randomized to treatment arm by restricted randomization and followed for the study period. While the arms were at the cluster level, outcomes were assessed both at the cluster level and at the individual level by taking random samples among those living in the study clusters.
Units Other Than Participants: Clusters
Groups:
- Community-wide Deworming (Intervention): Twice-yearly community-wide treatment delivered by drug distributors door to door for three years. All individuals above the age of 12 months (India/Benin) or 24 months of age (MalawI) who were not pregnant in the first trimester will receive a single dose of albendazole.
  The intervention followed delivery of the standard of care school-age-targeted deworming delivered annually (Benin/Malawi) or biannually (India) described below.
  Albendazole: All eligible individuals will receive a single dose of 400 mg albendazole.
- School-age-targeted Deworming (Control): Pre-school (pre-SAC) and school-age children (SAC) 1-14 years of age (Benin), 1-19 years of age (India) or 2-19 years of age (Malawi) were offered treatment in schools or community gatherings annually (Benin/Malawi) or twice-yearly (India) per standard of care national treatment guidelines for three years.
  Albendazole: All eligible individuals will receive a single dose of 400 mg albendazole.
Period: Overall Study
Arm/Group | Community-wide Deworming (Intervention) | School-age-targeted Deworming (Control)
Started | 177705; 60 Clusters | 179207; 60 Clusters
Completed (Assignment was at the study cluster level and individuals came in and out of the study due to in- and out-migration, births and deaths) | 119342; 60 Clusters (Assignment was at the study cluster level and individuals came in and out of the study due to in- and out-migration, births and deaths) | 116665; 60 Clusters (Assignment was at the study cluster level and individuals came in and out of the study due to in- and out-migration, births and deaths)
Not Completed | 58363; 0 Clusters | 62542; 0 Clusters

BASELINE CHARACTERISTICS:
Population: Censused population prior to the intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Community-wide Deworming (Intervention) | School-age-targeted Deworming (Control) | Total
Number analyzed (Participants) | 177705 | 180011 | 357716
Age, Customized [Count of Participants; unit: Participants]
  Age category: Infants (<1 year) | 4337 | 4396 | 8733
  Age category: Pre-school-age children (1-4 years) | 18491 | 18634 | 37125
  Age category: School-age children (5-14 years) | 42471 | 43062 | 85533
  Age category: Adults (15+ years) | 112284 | 113618 | 225902
  Age category: Unknown | 122 | 301 | 423
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 86233 | 87430 | 173663
  Sex: Female | 91466 | 92564 | 184030
  Sex: Other | 6 | 17 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Language: Majority language | 168000 | 169596 | 337596
  Language: Minority Language | 7334 | 8149 | 15483
  Language: Unknown | 2371 | 2266 | 4637
Region of Enrollment [Number; unit: participants]
  Benin | 48241 | 46728 | 94969
  Malawi | 61007 | 60811 | 121818
  India | 68457 | 72472 | 141929
Baseline STH prevalence: qPCR [Count of Participants; unit: Participants] — Population: Among participants who were censused and randomly selected into the baseline survey. each species is among total and therefore do not sum to totals
  Participants
    N. americanus: number analyzed (Participants) | 15119 | 14861 | 29980
    N. americanus | 2288 | 2214 | 4502
    A. lumbricoides: number analyzed (Participants) | 15119 | 14861 | 29980
    A. lumbricoides | 141 | 148 | 289
    A. duodenale: number analyzed (Participants) | 15119 | 14861 | 29980
    A. duodenale | 23 | 17 | 40
    T. trichiura: number analyzed (Participants) | 15119 | 14861 | 29980
    T. trichiura | 23 | 19 | 42
    Any STH species: number analyzed (Participants) | 15119 | 14861 | 29980
    Any STH species | 2444 | 2368 | 4812

OUTCOME MEASURES:

1. Secondary Outcome: N. Americanus Transmission Interruption - Pooled
Description: Prevalence of N. americanus infection ≤2% 24 months following the final round of mass drug administration with albendazole
Time Frame: 5 years (Three years of drug administration and two years of surveillance)
Population: The age- and sex-weighted prevalence of N. americanus was calculated at the cluster level and defined as transmission interruption if the bound of the one-side 95% confidence interval was <2%. The study cluster is a demarcated section of the study area (40 per country) with 1650+ individuals following local administrative boundaries.
Measure: Count of Units; unit: Study clusters
Units Other Than Participants: Study clusters
Arm/Group | Community-wide Deworming (Intervention) | School-age-targeted Deworming (Control)
Number analyzed (Participants) | 58554 | 58827
Number analyzed (Study clusters) | 60 | 60
Study clusters
  Transmission interruption | 12 | 6
  Did not achieve transmission interruption | 48 | 54

2. Secondary Outcome: Comparison of Arms - Pooled
Description: Individual-level soil-transmitted helminth species-specific endline quantitative PCR prevalence
Time Frame: 5 years (Three years of drug administration and two years of surveillance)
Population: The number of participants analyzed is the number surveyed and sampled at endline
Measure: Count of Participants; unit: Participants
Arm/Group | Community-wide Deworming (Intervention) | School-age-targeted Deworming (Control)
Number analyzed (Participants) | 58827 | 58554
Participants
  N. americanus (primary) | 3055 [0.36 to 0.48] | 7047
  A. duodenale | 20 [0.33 to 1.51] | 29
  A. lumbricoides | 152 [0.89 to 2.18] | 81
  T. trichiura | 22 [0.76 to 3.12] | 15
  Any STH species | 3243 [0.37 to 0.49] | 7153

3. Primary Outcome: Comparison of Arms - Benin
Description: Individual-level soil-transmitted helminth species-specific endline quantitative PCR prevalence
Time Frame: 5 years (Three years of drug administration and two years of surveillance)
Population: The number of participants analyzed is the number surveyed and sampled at endline
Measure: Count of Participants; unit: Participants
Arm/Group | Community-wide Deworming (Intervention) | School-age-targeted Deworming (Control)
Number analyzed (Participants) | 18490 | 18673
Participants
  N. americanus: N americanus | 322 | 748
  A duodenale: N americanus | 11 | 11
  A lumbricoides: N americanus | 123 | 59
  T trichiura: N americanus | 13 | 6
  Any STH species: N americanus | 467 | 819

4. Primary Outcome: Comparison of Arms - India
Description: Individual-level soil-transmitted helminth species-specific endline quantitative PCR prevalence
Time Frame: 5 years (Three years of drug administration and two years of surveillance)
Population: The number of participants analyzed is the number surveyed and sampled at endline
Measure: Count of Participants; unit: Participants
Arm/Group | Community-wide Deworming (Intervention) | School-age-targeted Deworming (Control)
Number analyzed (Participants) | 19894 | 19896
Participants
  N. americanus (primary) | 1906 [0.32 to 0.52] | 4310
  A. duodenale | 3 [0.17 to 4.94] | 3
  A. lumbricoides | 17 [0.81 to 5.29] | 7
  T. trichiura | 7 [0.34 to 2.67] | 5
  Any STH species | 1930 [0.33 to 0.52] | 4318 [na to na]

5. Primary Outcome: Comparison of Arms - Malawi
Description: Individual-level soil-transmitted helminth species-specific endline quantitative PCR prevalence
Time Frame: 5 years (Three years of drug administration and two years of surveillance)
Population: The number of participants analyzed is the number surveyed and sampled at endline
Measure: Count of Participants; unit: Participants
Arm/Group | Community-wide Deworming (Intervention) | School-age-targeted Deworming (Control)
Number analyzed (Participants) | 20170 | 20258
Participants
  N. americanus (primary) | 827 [0.34 to 0.46] | 1989 [na to na]
  A. duodenale | 6 [0.07 to 1.40] | 15 [na to na]
  A. lumbricoides | 12 [0.37 to 1.38] | 15 [na to na]
  T. trichiura | 2 [0.03 to 2.63] | 4 [na to na]
  Any STH species | 846 [0.35 to 0.47] | 2016 [na to na]

6. Primary Outcome: N. Americanus Transmission Interruption - Benin
Description: as for outcome 1
Time Frame: 5 years (Three years of drug administration and two years of surveillance)
Population: The age- and sex-weighted prevalence of N. americanus was calculated at the cluster level and defined as transmission interruption if the bound of the one-side 95% confidence interval was <2%.
Measure: Count of Units; unit: Study clusters
Units Other Than Participants: Study clusters
Arm/Group | Community-wide Deworming (Intervention) | School-age-targeted Deworming (Control)
Number analyzed (Participants) | 18490 | 18673
Number analyzed (Study clusters) | 20 | 20
Study clusters
  Transmission interruption | 11 | 6
  Did not achieve transmission interruption | 9 | 14

7. Primary Outcome: N. Americanus Transmission Interruption - India
Description: as for outcome 1
Time Frame: 5 years (Three years of drug administration and two years of surveillance)
Population: as for outcome 1
Measure: Count of Units; unit: Study clusters
Units Other Than Participants: Study clusters
Arm/Group | Community-wide Deworming (Intervention) | School-age-targeted Deworming (Control)
Number analyzed (Participants) | 19894 | 19896
Number analyzed (Study clusters) | 20 | 20
Study clusters
  Transmission interruption | 1 | 0
  Did not achieve transmission interruption | 19 | 20

8. Secondary Outcome: STH Transmission Interruption - Pooled
Description: Prevalence of STH infection ≤2% 24 months following the final round of mass drug administration with albendazole
Time Frame: 5 years (Three years of drug administration and two years of surveillance)
Population: The age- and sex-weighted prevalence of any STH species was calculated at the cluster level and defined as transmission interruption if the bound of the one-side 95% confidence interval was <2%.
Measure: Count of Units; unit: Study clusters
Units Other Than Participants: Study clusters
Arm/Group | Community-wide Deworming (Intervention) | School-age-targeted Deworming (Control)
Number analyzed (Participants) | 58554 | 58827
Number analyzed (Study clusters) | 60 | 60
Study clusters
  Transmission interruption | 9 | 5
  Did not achieve transmission interruption | 51 | 55

9. Secondary Outcome: STH Transmission Interruption - Benin
Description: Prevalence of STH infection ≤2% 24 months following the final round of mass drug administration with albendazole
Time Frame: 5 years (Three years of drug administration and two years of surveillance)
Population: as for outcome 8
Measure: Count of Units; unit: Study clusters
Units Other Than Participants: Study clusters
Arm/Group | Community-wide Deworming (Intervention) | School-age-targeted Deworming (Control)
Number analyzed (Participants) | 18490 | 18673
Number analyzed (Study clusters) | 20 | 20
Study clusters
  Transmission interruption | 9 | 5
  Did not achieve transmission interruption | 11 | 15

10. Secondary Outcome: STH Transmission Interruption - India
Description: Prevalence of STH infection ≤2% 24 months following the final round of mass drug administration with albendazole
Time Frame: 5 years (Three years of drug administration and two years of surveillance)
Population: The age- and sex-weighted prevalence of any STH was calculated at the cluster level and defined as transmission interruption if the bound of the one-side 95% confidence interval was <2%.
Measure: Count of Units; unit: Study clusters
Units Other Than Participants: Study clusters
Arm/Group | Community-wide Deworming (Intervention) | School-age-targeted Deworming (Control)
Number analyzed (Participants) | 19894 | 19896
Number analyzed (Study clusters) | 20 | 20
Study clusters
  Transmission interruption | 0 | 0
  Did not achieve transmission interruption | 20 | 20

11. Secondary Outcome: STH Transmission Interruption - Malawi
Description: Prevalence of STH infection ≤2% 24 months following the final round of mass drug administration with albendazole
Time Frame: 5 years (Three years of drug administration and two years of surveillance)
Population: as for outcome 8
Measure: Count of Units; unit: Study clusters
Units Other Than Participants: Study clusters
Arm/Group | Community-wide Deworming (Intervention) | School-age-targeted Deworming (Control)
Number analyzed (Participants) | 20170 | 20258
Number analyzed (Study clusters) | 20 | 20
Study clusters
  Transmission interruption | 0 | 0
  Did not achieve transmission interruption | 20 | 20

12. Primary Outcome: N. Americanus Transmission Interruption - Malawi
Description: as for outcome 1
Time Frame: 5 years (Three years of drug administration and two years of surveillance)
Population: as for outcome 1
Measure: Count of Units; unit: Study clusters
Units Other Than Participants: Study clusters
Arm/Group | Community-wide Deworming (Intervention) | School-age-targeted Deworming (Control)
Number analyzed (Participants) | 20170 | 20258
Number analyzed (Study clusters) | 20 | 20
Study clusters
  Transmission interruption | 0 | 0
  Did not achieve transmission interruption | 20 | 20

ADVERSE EVENTS:
Time Frame: 2 years, 9 months. Treatment with albendazole is known to be safe and billions of doses have been distributed over the previous decades. Therefore, a comparison between arms was not an objective of the study and adverse events were only collected to reduce the risk of harm to research subjects. Therefore, adverse events were passively ascertained during rounds of mass drug administration contacted the study staff and a study clinician reviewed and responded to adverse events.
Groups:
- Community-wide Deworming (Intervention): Twice-yearly community-wide treatment delivered by drug distributors door to door for three years. All individuals above the age of 12 months (India/Benin) or 24 months of age (Malawi) who were not pregnant in the first trimester will receive a single dose of albendazole.
  The intervention followed delivery of the standard of care school-age-targeted deworming delivered annually (Benin/Malawi) or biannually (India) described below.
  Albendazole: All eligible individuals will receive a single dose of 400 mg albendazole.
  NOTE: AEs were passively collected only in the intervention arm of the study as the government delivered the standard of care.
Arm/Group | Community-wide Deworming (Intervention)
All-Cause Mortality (participants affected / at risk) | 0/242344
Serious Adverse Events (participants affected / at risk) | 13/242344
Other Adverse Events (participants affected / at risk) | 0/242344
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Community-wide Deworming (Intervention) (N=242344)
Viral fever (Gastrointestinal disorders) | 1 (1) — Tested positive for Typhoid O&H and hospitalized
Acute gastroenteritis (Gastrointestinal disorders) | 3 (3) — Hospitalized
Fainting (General disorders) | 4 (4) — 4 cases of fainting following treatment with albendazole and praziquantel - all leading to hospitalization. Two were known epileptics and one also tested malaria positive
Fever / malaria (Infections and infestations) | 4 (4) — Hospitalization for severe malaria
Impacted bowel (Gastrointestinal disorders) | 1 (1) — Hospitalized

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT03014167/Prot_002.pdf
  • Statistical Analysis Plan (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT03014167/SAP_003.pdf